CLINICAL TRIAL: NCT06464575
Title: Prediction of a Structured Clinical Assessment by Patient Reported Outcomes and Machine Learning Algorithms: A Comparative Study
Brief Title: Comparison of Vocal Biomarkers for Depression and Anxiety to Formal Clinical Assessments
Status: Enrolling by invitation | Type: Observational
Sponsor: Ellipsis Health (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00070013
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-05

CONDITIONS: Depression/Anxiety
Keywords: Vocal biomarker; Depression; Anxiety; Structured clinical assessment
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

SUMMARY:
Participants will be recruited to complete self reported surveys normally used as standards of care for screening and monitoring depression and anxiety symptom severity, provide a voice sample composed of an answer to open ended questions and then be assessed by a mental health professional using structured and clinically validated assessment tools for depression and anxiety. Their voice will be analyzed by machine learning models that predict the severity of depression and anxiety symptoms. The models' performance will be compared to the clinician assessments and how that correlation compares to a similar comparison between the clinician assessments with the self reported surveys. It is hypothesized that the performance of the machine learning models in assessing the severity of depression and anxiety symptoms is no worse than the self reported surveys when both are compared to clinician assessments. It is also hypothesized that presence or absence of the diagnoses of Major Depressive Disorder and Generalized Anxiety Disorder can be predicted better than chance by the analysis of the participant's voice sample using machine learning models.

ELIGIBILITY:
Inclusion Criteria:

* Native speaker or conversant in English
* Access to smartphone or computer with microphone
* Provision of esigned and dated informed consent form
* Willingness to adhere to the study protocol
* To participate in the subsequent clinical interview portion of this study in addition to the above inclusion criteria, a participant must provide an evaluable and qualified voice sample.

Exclusion Criteria:

* Speech impairments or other conditions that impact their ability to speak clearly
* Under the influence of recreational drugs or alcohol
* Ill or experiencing heavy allergies or temporary conditions affecting respiration, voice, or speaking.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ~540 individuals aged 18 and above, of any gender, race, culture, ethnicity, sexual orientation or educational level residing anywhere in the United States.
Sampling Method: Non-Probability Sample
Enrollment: 540 (Estimated)
Dates: Start 2024-01-12 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome A | 4 days
  Extent of categorical agreement, measured in weighted kappa, between Ellipsis Health Software as a Medical Device severity of depression and clinician's rating of severity of depression.
Primary Outcome B | 4 days
  Extent of categorical agreement, measured in weighted kappa, between Ellipsis Health Software as a Medical Device severity of anxiety and clinician's rating of severity of anxiety.

SECONDARY OUTCOMES:
Secondary Outcome A | 4 days
  Extent of agreement of presence, measured in the Equal Error Rate on the Receiver Operating Characteristic curve, between Ellipsis Health Software aa a Medical Device detection of Major Depressive Disorder and clinician's assessment for the diagnosis of Major Depressive Disorder, as expressed as Sensitivity and Specificity.
Secondary Outcome B | 4 days
  Extent of agreement of presence, measured in the Equal Error Rate on the Receiver Operating Characteristic curve, between Ellipsis Health Software as a Medical Device detection of Generalized Anxiety Disorder and clinician's assessment for the diagnosis of Generalized Anxiety Disorder, as expressed as Sensitivity and Specificity.

CONTACTS AND LOCATIONS:
Locations (1):
- Ellipsis Health, San Francisco, California, United States